CLINICAL TRIAL: NCT00591773
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TAK-491 When Co-administered With Chlorthalidone in Subjects With Essential Hypertension
Brief Title: Efficacy and Safety of Azilsartan Medoxomil Co-Administered With Chlorthalidone in Participants With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-491-009; U1111-1113-9040 (Registry Identifier: WHO)
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
Keywords: Blood pressure; Blood pressure monitoring, ambulatory
MeSH Terms: conditions — Hypertension | interventions — azilsartan medoxomil; Chlorthalidone; azilsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Chlorthalidone 25 mg QD (Active Comparator)
  Interventions: Drug: Chlorthalidone

INTERVENTIONS:
Drug: Azilsartan medoxomil and chlorthalidone — Azilsartan medoxomil 40 mg, tablets, orally, once daily; azilsartan medoxomil 80 mg placebo-matching tablets, orally, once daily; and chlorthalidone 25 mg, tablets, orally, once daily for up to 6 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD
Drug: Azilsartan medoxomil and chlorthalidone — Azilsartan medoxomil 80 mg, tablets, orally, once daily; azilsartan medoxomil 40 mg placebo-matching tablets, orally, once daily and chlorthalidone 25 mg, tablets, orally, once daily for up to 6 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD
Drug: Chlorthalidone — Chlorthalidone 25 mg, tablets, orally, once daily; azilsartan medoxomil 80 mg placebo-matching tablets, orally, once daily and azilsartan medoxomil 40 mg placebo-matching tablets, orally, once daily for up to 6 weeks.
  Other Names: Thalitone
  Arms: Chlorthalidone 25 mg QD

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of azilsartan medoxomil, once daily (QD), co-administered with chlorthalidone in treating individuals with essential hypertension, compared to treatment with chlorthalidone alone.

DETAILED DESCRIPTION:
Hypertension affects approximately 50 million individuals in the United States. As the population ages, the prevalence of hypertension will continue to increase if broad and effective preventive measures are not implemented. According to the World Health Organization, hypertension is the most common attributable cause of preventable death in developed nations, as uncontrolled hypertension greatly increases the risk of cardiovascular disease, cerebrovascular disease, and renal failure. Despite the availability of antihypertensive treatments, hypertension remains inadequately controlled; only about one-third of patients continue to maintain control successfully.

TAK-491 (azilsartan medoxomil) is an angiotensin II receptor blocker that was shown to be a orally active antihypertensive agent with a prolonged duration of activity and good safety tolerability in a recent clinical study. Chlorthalidone is a thiazide-like diuretic that reduces blood pressure by decreasing intravascular volume through urinary salt and water excretion. By combining this action with azilsartan medoxomil, a greater reduction in blood pressure is expected than with either agent alone. For subjects requiring combination therapy, azilsartan medoxomil plus chlorthalidone offers a novel combination that may provide a more potent and safe combination for blood pressure reduction.

This study is being conducted to determine whether administration of azilsartan medoxomil in combination with chlorthalidone to subjects with uncontrolled hypertension is more effective in reducing blood pressure than chlorthalidone alone. This study is also being conducted to evaluate the safety and tolerability of azilsartan medoxomil combined with chlorthalidone.

Individuals who want to participate in this study will be required to provide written informed consent. Study participation is anticipated to be about 10 Weeks. Multiple procedures will occur at each visit which may include fasting, blood collection, urine collection, vital signs including sitting and standing blood pressure and pulse, body height and weight, physical examinations, electrocardiogram. Outside of the study center, participants will be required to wear an ambulatory blood pressure monitoring device at 24 hour intervals.

ELIGIBILITY:
Inclusion Criteria

1. Has essential hypertension (defined as sitting trough clinic systolic blood pressure between 160 and 190 mm Hg inclusive at Day minus 1 and 24-hour mean systolic blood pressure greater than or equal to 140 mm Hg and ≤ 180 mm Hg at Day 1).
2. Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
3. Has clinical laboratory evaluations (including clinical chemistry, hematology, and complete urinalysis) within the reference range for the testing laboratory or results that are deemed not clinically significant for inclusion into this study by the investigator.
4. Willing to discontinue current antihypertensive medications at the Screening Day minus 21 visit. If the subject is on amlodipine prior to screening, the subject is willing to discontinue this medication at Screening Day minus 28.

Exclusion Criteria

1. Has sitting trough clinic diastolic blood pressure greater than 119 mmHg at Day minus 1.
2. Has a baseline 24 hour ambulatory blood pressure monitor reading of insufficient quality.
3. Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication.
4. Recent history (within the last 6 months) of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
5. Clinically significant cardiac conduction defects (for example, 3rd degree atrioventricular block, left bundle branch block, sick sinus syndrome, atrial fibrillation).
6. Hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
7. The subject has secondary hypertension of any etiology.
8. Non-compliant (less than 70% or greater than 130%) with study medication
9. during the placebo run- in period.
10. Severe renal dysfunction or disease (based on calculated creatinine clearance less than 30 mL/min/1.73 m2) at Screening.
11. Known or suspected unilateral or bilateral renal artery stenosis.
12. History of drug abuse (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 2 alcoholic drinks per day) within the past 2 years.
13. Previous history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. (This criterion does not apply to those subjects with basal cell or Stage 1 squamous cell carcinoma of the skin.)
14. Type 1 or poorly controlled type 2 diabetes mellitus (glycosylated hemoglobin greater than 8.0%).
15. Hypo- or hyperkalemia (defined as serum potassium outside of the normal reference range of the central laboratory).
16. Alanine aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice.
17. Upper arm circumference less than 24 cm or greater than 42 cm.
18. Works night (3rd) shift (defined as 11PM [2300] to 7AM [0700]).
19. Currently is participating in another investigational study or has participated in an investigational study within 30 days prior to randomization.
20. Study site employee, or is an immediate family member ( ie, spouse, parent, child, sibling) of a study site employee who is involved in conduct of this study.
21. Any other serious disease or condition at Screening (or Randomization) that would compromise subject safety, might affect life expectancy, or make it difficult to successfully manage and follow the subject according to the protocol.
22. Randomized in a previous azilsartan medoxomil study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director Clinical Science, Study Director — Takeda
Locations (46):
- United States (46):
  - Huntsville, Alabama
  - Montgomery, Alabama
  - Buena Park, California
  - Huntington Beach, California
  - Long Beach, California
  - Mission Viejo, California
  - Roseville, California
  - Sacramento, California
  - Westlake Village, California
  - Coral Gables, Florida
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Miami, Florida
  - Auburn, Maine
  - Bingham Farms, Michigan
  - Troy, Michigan
  - Charlotte, North Carolina
  - Huntersville, North Carolina
  - Shelby, North Carolina
  - Akron, Ohio
  - Centerville, Ohio
  - Cincinnati, Ohio
  - Willoughby Hills, Ohio
  - Zanesville, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Tualatin, Oregon
  - Bensalem, Pennsylvania
  - Feasterville, Pennsylvania
  - Cranston, Rhode Island
  - Simpsonville, South Carolina
  - Kingsport, Tennessee
  - Corpus Christi, Texas
  - Houston, Texas
  - Pearland, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Arlington, Virginia
  - Burke, Virginia
  - Richmond, Virginia
  - Lakewood, Washington
  - Olympia, Washington
  - Port Orchard, Washington

REFERENCES:
- [Derived] Weber MA, Sever P, Juhasz A, Roberts A, Cao C. A randomized trial of the efficacy and safety of azilsartan medoxomil combined with chlorthalidone. J Renin Angiotensin Aldosterone Syst. 2018 Jul-Sep;19(3):1470320318795000. doi: 10.1177/1470320318795000. PMID 30175930

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 74 investigative sites in Argentina, Chile, Mexico, Peru and the United States from 07 September 2007 to 05 March 2009.
Pre-assignment Details: Participants with uncontrolled essential hypertension were enrolled in one of three, once-daily (QD) treatment groups.
Groups:
- Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD: Azilsartan medoxomil 40 mg, tablets, orally, once daily and chlorthalidone 25 mg, tablets, orally, once daily for up to 6 weeks.
- Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD: Azilsartan medoxomil 80 mg, tablets, orally, once daily and chlorthalidone 25 mg, tablets, orally, once daily for up to 6 weeks.
- Chlorthalidone 25 mg QD: Chlorthalidone 25 mg, tablets, orally, once daily for up to 6 weeks.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Started | 185 | 182 | 184
Completed | 169 | 158 | 168
Not Completed | 16 | 24 | 16
Not completed — Adverse Event | 9 | 9 | 6
Not completed — Protocol Violation | 2 | 3 | 0
Not completed — Lost to Follow-up | 1 | 4 | 1
Not completed — Withdrawal by Subject | 2 | 5 | 3
Not completed — Lack of Efficacy | 1 | 2 | 2
Not completed — Other | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD | Total
Number analyzed (Participants) | 185 | 182 | 184 | 551
Age Categorical [Number; unit: participants]
  <45 years | 21 | 15 | 16 | 52
  Between 45 and 64 years | 114 | 110 | 113 | 337
  ≥65 years | 50 | 57 | 55 | 162
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 88 | 82 | 266
  Male | 89 | 94 | 102 | 285

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 24-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 149 | 147 | 152
mmHg | -31.72 (0.966) | -31.30 (0.973) | -15.85 (0.957)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — Postbaseline P-value was from ANCOVA with terms for treatment (as a factor) and baseline value (as a covariate). Unadjusted p-value is presented. Overall 0.05 level of significance for multiple comparisons controlled using closed testing procedure; Mean Difference (Final Values) = -15.86, 95% CI 2-sided [-18.54 to -13.19]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -15.45, 95% CI 2-sided [-18.13 to -12.76]

2. Secondary Outcome: Change From Baseline in Mean Trough Clinic Sitting Systolic Blood Pressure.
Description: The change in mean trough clinic sitting systolic blood pressure measured at final visit or week 6 relative to baseline. Systolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 179 | 176 | 178
mmHg | -36.16 (1.226) | -34.44 (1.236) | -21.76 (1.229)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -14.40, 95% CI 2-sided [-17.81 to -10.99]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.68, 95% CI 2-sided [-16.10 to -9.25]

3. Secondary Outcome: Change From Baseline in the 24-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 149 | 147 | 152
mmHg | -18.28 (0.626) | -18.49 (0.630) | -7.99 (0.619)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — Postbaseline P-value was from ANCOVA with terms for treatment (as a factor) and baseline value (as a covariate). Unadjusted p-value is presented; Mean Difference (Final Values) = -10.29, 95% CI 2-sided [-12.02 to -8.56]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -10.49, 95% CI 2-sided [-12.23 to -8.76]

4. Secondary Outcome: Change From Baseline in Mean Trough Clinic Sitting Diastolic Blood Pressure.
Description: The change in mean trough clinic sitting diastolic blood pressure measured at final visit or week 6 relative to baseline. Diastolic blood pressure is the arithmetic mean of the 3 trough sitting diastolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 179 | 176 | 178
mmHg | -16.18 (0.717) | -15.98 (0.723) | -8.93 (0.719)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.25, 95% CI 2-sided [-9.25 to -5.25]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.05, 95% CI 2-sided [-9.06 to -5.05]

5. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 149 | 147 | 152
mmHg | -32.53 (0.996) | -31.97 (1.003) | -15.73 (0.988)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -16.80, 95% CI 2-sided [-19.56 to -14.04]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -16.24, 95% CI 2-sided [-19.01 to -13.47]

6. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 149 | 147 | 152
mmHg | -18.82 (0.665) | -18.99 (0.670) | -7.79 (0.659)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.02, 95% CI 2-sided [-12.86 to -9.18]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.20, 95% CI 2-sided [-13.04 to -9.35]

7. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 149 | 147 | 152
mmHg | -29.52 (1.080) | -29.43 (1.087) | -16.59 (1.069)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -12.93, 95% CI 2-sided [-15.92 to -9.94]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -12.84, 95% CI 2-sided [-15.83 to -9.84]

8. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 149 | 147 | 152
mmHg | -17.05 (0.714) | -17.06 (0.718) | -8.89 (0.707)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.16, 95% CI 2-sided [-10.14 to -6.19]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.17, 95% CI 2-sided [-10.15 to -6.19]

9. Secondary Outcome: Change From Baseline in the 12-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 12-hour mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 149 | 147 | 152
mmHg | -33.02 (1.039) | -32.45 (1.048) | -15.50 (1.031)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -17.52, 95% CI 2-sided [-20.39 to -14.64]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -16.95, 95% CI 2-sided [-19.84 to -14.05]

10. Secondary Outcome: Change From Baseline in the 12-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 12-hour mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 149 | 147 | 152
mmHg | -19.06 (0.706) | -19.20 (0.710) | -7.53 (0.698)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.54, 95% CI 2-sided [-13.49 to -9.59]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.68, 95% CI 2-sided [-13.64 to -9.72]

11. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 149 | 147 | 152
mmHg | -30.73 (1.118) | -30.16 (1.126) | -16.69 (1.108)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -14.04, 95% CI 2-sided [-17.13 to -10.94]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -13.48, 95% CI 2-sided [-16.58 to -10.37]

12. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 149 | 147 | 152
mmHg | -18.78 (0.804) | -19.04 (0.810) | -9.36 (0.797)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -9.42, 95% CI 2-sided [-11.65 to -7.20]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -9.69, 95% CI 2-sided [-11.92 to -7.46]

13. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Systolic Blood Pressure Response, Defined as < 140 mm Hg and/or Reduction From Baseline ≥ 20 mm Hg
Description: Percentage of participants who achieve a clinic systolic blood pressure response measured at week 6, defined as less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Systolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 179 | 176 | 178
percentage of participants | 87.7 | 84.1 | 63.5
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for response criteria for systolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic systolic blood pressure as a covariate. The unadjusted p-value is presented; Odds Ratio (OR) = 4.09, 95% CI 2-sided [2.38 to 7.03]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.03, 95% CI 2-sided [1.82 to 5.03]

14. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Diastolic Blood Pressure Response, Defined as < 90 mm Hg and/or Reduction From Baseline ≥ 10 mm Hg
Description: Percentage of participants who achieve a clinic diastolic blood pressure response measured at week 6 , defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg. Diastolic blood pressure is the arithmetic mean of the 3 trough sitting diastolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 179 | 176 | 178
percentage of participants | 92.7 | 90.3 | 78.1
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for response criteria for diastolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic diastolic blood pressure as a covariate. The unadjusted p-value is presented; Odds Ratio (OR) = 3.72, 95% CI 2-sided [1.90 to 7.27]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p = 0.002, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Odds Ratio (OR) = 2.70, 95% CI 2-sided [1.46 to 5.00]

15. Secondary Outcome: Percentage of Participants Who Achieve Both a Clinic Diastolic and Systolic Blood Pressure Response.
Description: Percentage of participants who achieve both a clinic diastolic and systolic blood pressure response measured at week 6, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg AND less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Diastolic and systolic blood pressure is based on the arithmetic mean of the 3 sitting blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Number analyzed (Participants) | 179 | 176 | 178
percentage of participants | 84.9 | 80.7 | 58.4
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for joint response criteria for systolic blood pressure and diastolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic systolic blood pressure as a covariate. The unadjusted p-value is presented; Odds Ratio (OR) = 4.00, 95% CI 2-sided [2.41 to 6.64]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD vs Chlorthalidone 25 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 2.96, 95% CI 2-sided [1.83 to 4.79]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD | Chlorthalidone 25 mg QD
Serious Adverse Events (participants affected / at risk) | 3/184 | 3/182 | 1/181
Other Adverse Events (participants affected / at risk) | 34/184 | 31/182 | 29/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD (N=184) | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD (N=182) | Chlorthalidone 25 mg QD (N=181)
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Heart rate decreased (Investigations) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg QD and Chlorthalidone 25 mg QD (N=184) | Azilsartan Medoxomil 80 mg QD and Chlorthalidone 25 mg QD (N=182) | Chlorthalidone 25 mg QD (N=181)
Plasminogen activator inhibitor increased (Investigations) | 12 | 4 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4 | 11
Dizziness (Nervous system disorders) | 16 | 19 | 6
Headache (Nervous system disorders) | 8 | 9 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.